CLINICAL TRIAL: NCT00981630
Title: Randomised, Double-blind, Placebo Controlled Phase II, Dose-ranging Study of the Safety, Tolerability and Immunogenicity of Live Attenuated ChimeriVax™-JE Vaccine (Lyophilised)
Brief Title: Study of Live Attenuated ChimeriVax™-Japanese Encephalitis Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-007
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; ChimeriVax™-JE Vaccine; Adult
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ChimeriVax™-JE Dose Level 1 (Experimental): Participants received ChimeriVax™-JE (Japanese Encephalitis) a dose of 3.0 log10 Plaque-forming units (PFU) on Day 0.
  Interventions: Biological: Live attenuated Japanese encephalitis virus
- ChimeriVax™-JE Dose Level 2 (Experimental): Participants received ChimeriVax™-JE a dose of 4.0 log10 PFU on Day 0.
  Interventions: Biological: Live attenuated Japanese encephalitis virus
- ChimeriVax™-JE Dose Level 3 (Experimental): Participants received ChimeriVax™-JE a dose of 5.0 log10 PFU on Day 0.
  Interventions: Biological: Live attenuated Japanese encephalitis virus
- Placebo (Placebo Comparator): Participants received ChimeriVax diluent, 0.5 mL on Day 0.
  Interventions: Biological: ChimeriVax™ diluent (Placebo)

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis virus — 0.5 mL,Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: ChimeriVax™-JE Dose Level 1
Biological: Live attenuated Japanese encephalitis virus — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: ChimeriVax™-JE Dose Level 2
Biological: Live attenuated Japanese encephalitis virus — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™-JE
  Arms: ChimeriVax™-JE Dose Level 3
Biological: ChimeriVax™ diluent (Placebo) — 0.5 mL, Subcutaneous
  Other Names: Paricipants received a dose of ChimeriVax™ diluent at Day 0.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of a new formulation of lyophilised ChimeriVax™-JE, given at three dose levels, compared with placebo.

Primary Objectives:

Safety:

* To obtain safety and tolerability data for a single subcutaneous vaccination with ChimeriVax™-JE, at three dose levels, in healthy adult volunteers (18-49 years old).

Immunogenicity:

* To obtain data on the antibody response to a single subcutaneous vaccination with ChimeriVax™-JE, at three dose levels, in healthy adult volunteers without prior Japanese encephalitis immunity.
* To assess the durability of immune response up to 12 months following a single subcutaneous vaccination with ChimeriVax™-JE, at three dose levels.

DETAILED DESCRIPTION:
All participants will received a single dose of study vaccine, ChimeriVax™-JE or placebo on Day 0. The double-blind treatment phase will last 30 days, with follow-up visits at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria :

* All aspects of the protocol explained and written informed consent obtained from the participant.
* Aged ≥18 to < 49 years.
* In good general health, without significant medical history, physical examination findings, or clinically significant abnormal laboratory results.
* Participant must be available for the study duration, including all planned follow-up visits.
* Participant must agree to take the following precautions to avoid insect bites for 7 days following vaccination by using N,N-diethyl-meta-toluamide (DEET)-containing insect repellent, where appropriate.
* For female participants: Negative pregnancy tests at Screening and Day 0, in conjunction with a menstrual and contraceptive history indicating a low probability of pregnancy in the opinion of the physician. Females of childbearing potential will be required to be correctly using an efficacious hormonal method of contraception or intrauterine device for at least 1 month before randomisation and during the on-study phase to Day 30. Barrier methods of contraception will not be considered acceptable for study entry. Female participants of child-bearing potential will sign an agreement that contraception will be correctly practised during the specified periods and will specify the method used. Female participants unable to become pregnant must have this documented (e.g., tubal ligation, hysterectomy or postmenopausal [at least one year since last menstrual period]).

Exclusion Criteria :

* A history of vaccination or infection to Japanese encephalitis (JE) or yellow fever (YF) or other flaviviruses (including Japanese encephalitis, tick-borne encephalitis, St Louis encephalitis, West Nile virus, dengue fever, Murray Valley encephalitis). Previous vaccination will be determined by history (interview of subject).
* Previous or current military service.
* History of residence in or travel to flavivirus endemic areas in the tropics (Cape York region of Northern Queensland, India, Southeast Asia, Central America, Caribbean or South America) for periods of 4 weeks or more.
* Known or suspected immunodeficiency (e.g., human immunodeficiency virus [HIV] infection, primary immunodeficiency disorder, leukemia, lymphoma), use of immunosuppressive or antineoplastic drugs (corticosteroids > 10 mg prednisone, or equivalent, in the last three months or during the trial (up to Day 30).
* History of thymoma, thymic surgery (removal) or myasthenia gravis.
* Clinically significant abnormalities on laboratory assessment (i.e., meeting the mild, moderate or severe criteria described in the toxicity gradings for laboratory values).
* Anaphylaxis or other serious adverse reactions characterised by urticaria or angioedema to foods, hymenoptera (bee family) stings, or drugs (including vaccines).
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within six months of the Screening Visit or up to Day 30.
* Administration of another vaccine or antiviral within 30 days preceding the screening visit or up to Day 30 (these subjects will be rescheduled for vaccination at a later date).
* Physical examination indicating any clinically significant medical condition.
* Body temperature > 38.1°C (100.6°F) or acute illness within 3 days prior to inoculation (participant may be rescheduled).
* Intention to travel out of the area prior to the study visit on Day 30.
* Seropositive to hepatitis C virus or HIV or positive for Hepatitis B Surface Antigen.
* Lactation or intended pregnancy in female subjects.
* Excessive alcohol consumption, drug abuse, significant psychiatric illness.
* A known or suspected physiological or structural condition that compromises the integrity of the blood-brain barrier (e.g., significant hypertensive cerebrovascular disease, trauma, ischaemia, infection, inflammation of the brain).
* Intention to increase normal exercise routine, participate in contact sports or strenuous weight lifting or to initiate vigorous exercise from Screening until after Day 30.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Australia (2):
  - Herston, Queensland
  - Adelaide, South Australia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 01 December 2004 to 31 January 2005 at 2 clinical centers in Australia.
Pre-assignment Details: A total of 128 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- ChimeriVax™-JE 3 log10 PFU: All participants received a single dose of ChimeriVax™-JE 3 log10 Plaque-forming units (PFU) vaccine on Day 0.
- ChimeriVax™-JE 4 log10 PFU: All participants received a single dose of ChimeriVax™-JE 4 log10 Plaque-forming units (PFU) vaccine on Day 0.
- ChimeriVax™-JE 5 log10 PFU: All participants received a single dose of ChimeriVax™-JE 5 log10 Plaque-forming units (PFU) vaccine on Day 0
- Placebo: All participants received a single dose of Placebo (diluent) on Day 0.
Period: Overall Study
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Started | 32 | 32 | 32 | 32
Completed | 32 | 32 | 32 | 32
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 32 | 32 | 128
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (7.62) | 26.7 (9.17) | 27.4 (8.31) | 29.4 (8.43) | 28.2 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 15 | 16 | 64
  Male | 17 | 14 | 17 | 16 | 64
Region of Enrollment [Number; unit: Participants]
  Australia | 32 | 32 | 32 | 32 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Seroconverted to the Respective Homologous JE Vaccine Strain, 28 Days After Completion of the Primary Immunization Schedule With One of 3 Doses of ChimeriVax™-JE Vaccine or A Placebo
Description: Antibodies were measured using 50% plaque reduction neutralization test (PRNT50) for measurement of neutralizing antibodies against homologous ChimeriVax™-JE and wild type JE virus strains. Seroconversion was defined as a titer ≥ 1:20 at post vaccination timepoints for subjects who were seronegative at baseline, or ≥ 4 fold rise from baseline.
Time Frame: Day 11 and Day 30 post-vaccination
Population: Seroconversion was assessed in all participants who were negative for homologous and all wild type JE antibodies at Day 0 and had no protocol violations that might have interfered with evaluation of primary criterion.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 32
Participants
  Day 11 | 1 | 10 | 8 | 0
  Day 30 | 31 | 30 | 29 | 1

2. Primary Outcome: Number of Participants Who Seroconverted to Wild Type JE Virus Strains After Primary Immunization Schedule With One of 3 Doses of ChimeriVax™-JE Vaccine or a Placebo
Description: Antibodies were measured using 50% plaque reduction neutralization test (PRNT50) for measurement of neutralizing antibodies against homologous ChimeriVax™-JE and wild type JE virus strains. Seroconversion was defined as a titer ≥ 1:20 at post vaccination time points for subjects who were seronegative at baseline, or ≥ 4 fold rise from baseline.
Time Frame: Day 30 post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 32
Participants
  Genotype I | 31 | 28 | 30 | 1
  Genotype II | 25 | 25 | 25 | 0
  Genotype III Beijing | 31 | 30 | 30 | 1
  Genotype III P3 | 30 | 29 | 29 | 0
  Genotype III Nakayama | 31 | 27 | 27 | 1
  Genotype IV | 25 | 28 | 26 | 0

3. Primary Outcome: Number of Participants Reporting Solicited Local Injection Site and Treatment Related Adverse Events Post Vaccination With One of 3 Doses of ChimeriVax™-JE Vaccine or Placebo
Description: Local Injection Site Adverse Events (AEs): Pain, Erythema, Reaction, Hemorrhage, Induration, Paresthesia. Treatment Related Systemic AEs: Fever, Chills, Malaise, Fatigue, Headache, Myalgia, Arthralgia, Nausea, Vomiting, Diarrhea, Rash. Other AEs as reported spontaneously.
Time Frame: Day 0 (post-vaccination) up to Day 30 post-vaccination
Population: Adverse events were assessed in all randomized participants who received one injection of study treatment, according to the treatment actually received (Safety Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants
  Injection Site Pain | 1 | 2 | 4 | 2
  Injection Site Erythema | 2 | 2 | 4 | 0
  Injection Site Reaction | 1 | 0 | 0 | 1
  Injection Site Hemorrhage | 0 | 3 | 2 | 1
  Injection Site Induration | 0 | 1 | 0 | 0
  Injection Site Paresthesia | 0 | 1 | 2 | 1
  Headache | 11 | 9 | 13 | 11
  Lethargy | 0 | 4 | 2 | 2
  Fatigue | 6 | 11 | 7 | 6
  Malaise | 4 | 7 | 5 | 2
  Feeling Hot | 0 | 2 | 2 | 3
  Chills | 0 | 2 | 2 | 1
  Myalgia | 2 | 6 | 9 | 2
  Arthralgia | 0 | 2 | 2 | 0
  Nausea | 0 | 6 | 3 | 2
  Diarrhea | 0 | 1 | 4 | 2
  Abdominal Pain | 0 | 4 | 1 | 1
  Pharyngitis | 2 | 3 | 3 | 4
  Diarrhea Infectious | 0 | 2 | 0 | 0
  Rhinorrhea | 2 | 1 | 0 | 1
  Pruritus | 0 | 1 | 1 | 2
  Neutropenia | 4 | 0 | 2 | 0
  Leukopenia | 2 | 3 | 0 | 0
  Lymphadenopathy | 0 | 2 | 1 | 1

4. Secondary Outcome: Geometric Mean Titers to Japanese Encephalitis (Homologous Virus) Following Primary Immunization Schedule With One of 3 Doses of ChimeriVax™-JE Vaccine or a Placebo
Description: Antibodies were measured using 50% plaque reduction neutralization test (PRNT50) for measurement of neutralizing antibodies against homologous ChimeriVax™-JE virus strains.
Time Frame: Day 11 and Day 30 post-vaccination
Population: Geometric Mean Titers were assessed in all participants who were negative for homologous and all wild type JE antibodies at Day 0 and had no protocol violations that might have interfered with evaluation of primary criterion (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 32
Titers
  Day 11 | 5.2 [4.8 to 5.7] | 11.4 [7.0 to 18.7] | 10.2 [6.3 to 16.5] | 5.0 [5.0 to 5.0]
  Day 30 | 1829.6 [916.6 to 3651.9] | 2151.5 [994.1 to 4656.8] | 1956.5 [913.4 to 4190.9] | 5.8 [4.3 to 7.9]

5. Secondary Outcome: Geometric Mean Titers to Japanese Encephalitis (Wild Type JE Virus Strains) Following Primary Immunization Schedule With One of 3 Doses of ChimeriVax™-JE Vaccine or a Placebo
Description: The Japanese Encephalitis (Wild Type JE Virus Strains) antibodies were measured using PRNT50 for measurement of neutralizing antibodies against homologous ChimeriVax™-JE and wild type JE virus strains.
Time Frame: Day 30 post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 32
Titers
  Genotype I | 208.6 [134.8 to 322.9] | 193.0 [109.4 to 340.5] | 188.3 [122.1 to 290.6] | 5.3 [4.7 to 5.9]
  Genotype II | 50.9 [33.8 to 76.5] | 69.2 [41.4 to 115.7] | 49.6 [32.2 to 76.3] | 5.0 [5.0 to 5.0]
  Genotype III (Beijing) | 232.6 [147.0 to 368.1] | 162.3 [91.0 to 289.6] | 253.4 [152.8 to 420.1] | 5.4 [4.7 to 6.2]
  Genotype III (P3) | 223.6 [147.3 to 339.4] | 238.7 [125.7 to 453.2] | 315.5 [182.0 to 547.0] | 5.3 [4.9 to 5.9]
  Genotype III (Nakayama) | 192.3 [127.3 to 290.6] | 180.6 [95.4 to 341.7] | 155.0 [83.6 to 287.3] | 5.6 [4.7 to 6.6]
  Genotype IV | 70.4 [42.4 to 117.1] | 80.4 [47.1 to 137.2] | 67.1 [41.3 to 108.8] | 5.0 [5.0 to 5.0]

6. Secondary Outcome: Participants With Japanese Encephalitis (Homologous Virus) Seropositivity Over Time Following Primary Immunization Schedule With One of 3 Doses of ChimeriVax™-JE Vaccine or Placebo
Description: Antibodies were measured using 50% plaque reduction neutralization test (PRNT50) for measurement of neutralizing antibodies against homologous ChimeriVax™-JE virus strains. Seropositivity was defined as a titer < 1:10.
Time Frame: Day 30 up to 12 months post-vaccination
Population: Seropositivity was assessed in all participants who were negative for homologous and all wild type JE antibodies at Day 0 and had no protocol violations that might have interfered with evaluation of primary criterion (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 32
Participants
  Day 30 [N = 31; 32; 31; 32] | 31 | 30 | 29 | 1
  Month 6 [N = 31; 30; 28; 32] | 30 | 28 | 27 | 0
  Month 12 [N = 31; 30; 30; 29] | 27 | 26 | 29 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to Month 12 post-vaccination.
Arm/Group | ChimeriVax™-JE 3 log10 PFU | ChimeriVax™-JE 4 log10 PFU | ChimeriVax™-JE 5 log10 PFU | Placebo
Serious Adverse Events (participants affected / at risk) | 2/32 | 1/32 | 0/32 | 2/32
Other Adverse Events (participants affected / at risk) | 16/32 | 16/32 | 16/32 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax™-JE 3 log10 PFU (N=32) | ChimeriVax™-JE 4 log10 PFU (N=32) | ChimeriVax™-JE 5 log10 PFU (N=32) | Placebo (N=32)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ChimeriVax™-JE 3 log10 PFU (N=32) | ChimeriVax™-JE 4 log10 PFU (N=32) | ChimeriVax™-JE 5 log10 PFU (N=32) | Placebo (N=32)
Headache (Nervous system disorders) | 16 | 16 | 16 | 17
Lethargy (Nervous system disorders) | 0 | 4 | 2 | 2
Fatigue (General disorders) | 6 | 16 | 10 | 7
Injection Site Pain (General disorders) | 1 | 2 | 4 | 2
Injection Site Erythema (General disorders) | 2 | 2 | 4 | 0
Injection Site Hemorrhage (General disorders) | 0 | 3 | 2 | 1
Injection Site Paresthesia (General disorders) | 0 | 1 | 2 | 1
Malaise (General disorders) | 7 | 7 | 6 | 7
Feeling Hot (General disorders) | 0 | 2 | 2 | 3
Chills (General disorders) | 0 | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 10 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 6 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 3 | 3 | 5
Diarrhea Infectious (Infections and infestations) | 0 | 2 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 1 | 1 | 2
Thrombocytopena (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 1 | 3
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Blood creatinine phosphokinase increased (Investigations) | 2 | 2 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 3 | 2 | 1
Bradycardia (Cardiac disorders) | 1 | 2 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.